CLINICAL TRIAL: NCT07212114
Title: A Randomized, Double-blind, Active Controlled, Single-center Study to Evaluate the Efficacy of EXPAREL vs. Bupivacaine HCl Administered as Combined Sciatic (in the Popliteal Fossa) and Saphenous (in the Adductor Canal) Nerve Blocks for Postsurgical Analgesia in Subjects Undergoing Total Ankle Arthroplasty
Brief Title: Efficacy of EXPAREL vs. Bupivacaine
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Principal Investigator, Sameh Labib, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00008684
Record Dates: First submitted 2025-09-02; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Total Ankle Arthroplasty; Postsurgical Analgesia
Keywords: Pain management; Postsurgical Analgesia; Bupivacaine; EXPAREL
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Admix (Experimental): EXPAREL admixed with 0.25% bupivacaine HCl Total volume (50 mL) will be split such that 30 mL will be administered as the sciatic nerve block (in the popliteal fossa) and 20 mL will be administered as the saphenous nerve block (in the adductor canal)
  Interventions: Drug: EXPAREL; Drug: 0.25% bupivacaine (HCl): 30 ml
- Reference (Experimental): Bupivacaine HCl arm Total volume (50 mL) will be split such that 30 mL will be administered as the sciatic nerve block (in the popliteal fossa) and 20 mL will be administered as the saphenous nerve block (in the adductor canal)
  Interventions: Drug: 0.25% bupivacaine (HCl): 50 ml

INTERVENTIONS:
Drug: EXPAREL — EXPAREL (bupivacaine liposome injectable suspension) is formulated as a sterile, non-pyrogenic, white to off-white, preservative-free homogenous suspension of bupivacaine encapsulated into multivesicular liposomes (pMVL drug delivery system). For this study, EXPAREL will be provided in 20 mL (266 mg) EXPAREL single-use, clear glass vials.
  Other Names: bupivacaine liposome injectable suspension
  Arms: Admix
Drug: 0.25% bupivacaine (HCl): 50 ml — The reference product is 50 mL (125 mg) 0.25% bupivacaine HCl administered via a combined sciatic (in the popliteal fossa) and saphenous nerve block (in the adductor canal)
  Arms: Reference
Drug: 0.25% bupivacaine (HCl): 30 ml — EXPAREL admixed with 30 mL (75 mg) 0.25% bupivacaine HCl
  Arms: Admix

SUMMARY:
The goal of this clinical study is to learn about pain management strategies in subjects undergoing total ankle replacement. arthroplasty surgery The primary objective is to compare the magnitude of the analgesic effect following a single dose injection of EXPAREL vs. 0.25% bupivacaine (HCl).

Secondary objectives are to:

Compare the total opioid consumption (in oral morphine equivalents) from 0 to 96 hours following a single dose injection of EXPAREL vs. 0.25% bupivacaine HCl

* Compare the time to first opioid consumption following a single dose injection of EXPAREL vs. 0.25% bupivacaine HCl
* Assess the safety of EXPAREL vs. 0.25% bupivacaine HCl
* Evaluate subject satisfaction with pain management following a single-dose injection of EXPAREL vs. 0.25% bupivacaine hydrochloride (HCl)
* Compare clinical performance from Preoperative status to 3- and 12- months postoperatively

DETAILED DESCRIPTION:
EXPAREL® is a long-acting local anesthetic specifically developed to provide extended postsurgical pain relief from a single-dose administration, thereby reducing or eliminating the need for indwelling catheters and minimizing reliance on supplemental opioid medications. It is currently indicated for single-dose infiltration to produce local analgesia in patients aged 6 years and older, as well as for regional analgesia via interscalene brachial plexus, sciatic (in the popliteal fossa), and adductor canal nerve blocks in adults. Pain following surgery is common, often peaking in the initial postoperative days, and if inadequately managed, it can delay healing, impair mobilization, prolong hospital stays, and increase the risk of complications and healthcare costs. Despite the prevalence of multimodal analgesic strategies-including the use of local anesthetics and systemic opioids-opioids remain a mainstay for moderate to severe postsurgical pain. However, their use is often limited by adverse effects such as respiratory depression, nausea, vomiting, pruritus, constipation, somnolence, and urinary retention. These complications not only reduce patient satisfaction and recovery but also increase medical intervention and resource use, making opioid-sparing alternatives clinically and economically attractive.

EXPAREL addresses this need by leveraging a proprietary multivesicular liposome (pMVL) drug delivery system that encapsulates bupivacaine at a concentration of 13.3 mg/mL within microscopic spherical vesicles. These vesicles-composed of naturally occurring or bioanalogous lipids-release bupivacaine gradually over time through lipid membrane reorganization and diffusion, thereby extending its duration of action well beyond the 6-8 hours typical of conventional bupivacaine formulations. The liposomal technology used in EXPAREL is based on the same pMVL platform found in the FDA-approved product DepoCyt®, though EXPAREL's lipid formulation has been modified for local anesthetic use. Since its initial FDA approval in 2011 for surgical site infiltration and the subsequent expansion of its indications in 2018 to include various nerve blocks, EXPAREL has been administered to approximately 14 million patients in the U.S., highlighting its growing adoption in clinical practice.

The rationale for the current study stems from the need to optimize postsurgical pain control in patients undergoing total ankle arthroplasty, a procedure associated with significant postoperative pain. This randomized, double-blind, active-controlled, single-center trial will evaluate the efficacy of EXPAREL when used in combination with bupivacaine HCl as part of a combined sciatic (popliteal fossa) and saphenous (adductor canal) nerve block regimen. Specifically, the intervention group will receive 20 mL EXPAREL (266 mg) admixed with 20 mL of 0.25% bupivacaine HCl (50 mg), while the control group will receive 40 mL of 0.25% bupivacaine HCl (100 mg), with each agent administered in equal volumes to the respective nerve sites. The objective is to determine whether the EXPAREL-based regimen provides more effective and longer-lasting analgesia compared to bupivacaine HCl alone, thereby enhancing recovery, reducing opioid consumption, and improving overall patient outcomes in a high-pain surgical population.

ELIGIBILITY:
Inclusion Criteria:

* Indicated to undergo unilateral total ankle arthroplasty
* American Society of Anesthesiologists (ASA) physical status 1, 2, or 3
* Able to provide informed consent, adhere to the study schedule, and complete all study assessments
* Body Mass Index (BMI) ≥18 and ≤40 kg/m2

Exclusion Criteria:

* Allergy, hypersensitivity, intolerance, or contraindication to any of the study medications for which an alternative is not named in the protocol (e.g., amide-type local anesthetics, opioids, bupivacaine HCl, NSAIDs)
* Concurrent painful physical condition that may require analgesic treatment (such as long-term, consistent use of opioids) in the post-dosing period for pain, and which, in the Investigator's opinion, may confound the post-dosing assessments
* History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years
* Uncontrolled anxiety, schizophrenia, or other psychiatric disorder that, in the opinion of the Investigator, could interfere with study assessments or compliance
* Currently pregnant, nursing, or planning to become pregnant during the study
* History of contralateral ankle arthroplasty within 1 year
* Subjects that require ankle arthroplasty due to failed prior ankle arthrodesis
* Subjects with avascular necrosis of the talus
* Subjects undergoing revision total ankle arthroplasty
* Clinically significant medical disease that, in the opinion of the Investigator, would make participation in a clinical study inappropriate. This includes diabetic neuropathy, coagulation or bleeding disorders, severe peripheral vascular disease, renal insufficiency, hepatic dysfunction or other conditions that would constitute a contraindication to participation in the study
* Chronic opioid use within 30 days before randomization (average ≥30 oral morphine equivalents/day
* Prisoners
* Cognitive impairment or impaired decision-making capacity
* Inability to communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Magnitude of the analgesic effect | Perioperative (Upon arrival in the PACU (±5 min), Postoperative (At PACU discharge (±5 min)), Every 6 hours from the end of surgery until health care facility discharge up to 96h
  To measure this, the Area under the curve (AUC) of the Numeric Rating Scale (NRS) for both groups will be compared.
  The subjects will be asked to rate their worst or average pain on a scale of 0 (no pain) - 10 (worst possible pain) on numerous time points, starting upon arrival in the Post-Anesthesia Care Unit (PACU)

SECONDARY OUTCOMES:
Total opioid consumption | Baseline (Hour 0), 96 hours post surgery
  Compare the total opioid consumption (in oral morphine equivalents) from 0 to 96 hours following a single dose injection of EXPAREL vs. 0.25% bupivacaine HCl
Time to first opioid consumption | Baseline (Hour 0), 96 hours post surgery
  Compare the time to first opioid consumption in oral morphine equivalents (OMED) following a single dose injection of EXPAREL vs. 0.25% bupivacaine HCl
Patient safety | Baseline (Hour 0), Day 14 post op
  Safety of EXPAREL vs. 0.25% bupivacaine HCl will be assessed by the Incidence of treatment-emergent Adverse Events and Serious AEs from the start of the nerve block procedure through Post op day (POD) 14
Subject satisfaction | Within 96 hours post op
  Subject satisfaction with pain management following the intervention in both groups will be assessed using a Subject Satisfaction Questionnaire. This consists of a single question asking participants to rate their satisfaction with pain management outcomes on a scale from 0 to 10, where 0 indicates 'extremely dissatisfied' and 10 indicates 'extremely satisfied
Pain intensity: Numeric Rating Scale (NRS) Short term | Every 6 hours from the end of surgery until health care facility discharge up to 96h
  Pain intensity will be measured using the 11-point NRS. The subject will be asked to rate their worst or average pain on a scale of 0 (no pain) to 10 (worst possible pain) in the operative ankle.
  This will be measured up to 96 hours post op.
Pain intensity: Numeric Rating Scale (NRS) : post discharge | Twice daily from the day of discharge upto Day 7 days post discharge
  Pain intensity will be measured using the 11-point NRS. The subject will be asked to rate their worst or average pain on a scale of 0 (no pain) to 10 (worst possible pain) in the operative ankle.
  Twice daily from the day 1 of discharge up to Day 7 post-discharge
Pain intensity: Numeric Rating Scale (NRS): Long term | Twice daily from the day 7 of discharge upto Day 14 post discharge
  Pain intensity will be measured using the 11-point NRS. The subject will be asked to rate their worst or average pain on a scale of 0 (no pain) to 10 (worst possible pain) in the operative ankle.
  Twice daily from day 7 of discharge up to 14 days post-discharge
Clinical Performance: SF-12 | Preoperative, 3 months post op, 12 months post op
  Scoring the SF-12 Health Survey involves calculating two key summary scores: the Physical Component Summary (PCS-12) and the Mental Component Summary (MCS-12). These scores reflect a person's overall physical and mental health status, respectively, and are derived from responses to 12 questions covering eight health domains.
  Standardized Scores: Both PCS-12 and MCS-12 are scored on a scale where:
  * A score above 50 indicates better-than-average health.
  * A score below 50 suggests worse-than-average health.
Clinical Performance: Ankle Osteoarthritis Score | Preoperative, 3 months post op, 12 months post op
  The Ankle Osteoarthritis Score (AOS) is a patient-reported outcome measure designed to assess pain and functional limitations caused by ankle osteoarthritis. It uses a series of visual analogue scales (VAS) where patients rate their pain and difficulty performing daily activities over the past week.
  Pain Subscale: Assesses ankle pain in various situations (e.g., walking barefoot, standing with shoes, end of day).
  Disability Subscale: Evaluates difficulty with activities like walking on uneven ground, climbing stairs, or running.
  Each item is rated on a 100 mm VAS line.
  * Scores range from 0 (no pain/difficulty) to 100 (worst imaginable pain or complete inability).
  * Subscale scores are calculated by averaging the responses within each category.
  * The total AOS score is the average of the pain and disability subscale scores.

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Labib, MD, FAOA, Principal Investigator — Emory University
Locations (1):
- Emory University Orthopaedic Hospital Musculoskeletal Institute (MSK), Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified participant data will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be made available beginning 6 months after publication of the primary study results